CLINICAL TRIAL: NCT02623894
Title: Influence of Different Risk Factors in Vascular Accelerated Aging. A Cross-sectional, Descriptive Observational Study (EVA Study)
Brief Title: Influence of Different Risk Factors in Vascular Accelerated Aging (EVA Study)
Status: Completed | Type: Observational
Sponsor: Fundacion para la Investigacion y Formacion en Ciencias de la Salud (Other)
Collaborators: Castilla-León Health Service (Other)
Responsible Party: Sponsor
Other Study IDs: GRS 1193/B/15
Record Dates: First submitted 2015-11-23; First posted 2015-12-08 (Estimated); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Healthy
Keywords: Vascular aging.; Arterial stiffness.; Lifestyles.; Vascular structure.; Telomere length,; Psychological factors.; Inflammatory factors.; Oxidative stress

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — Fasting plasma glucose, creatinine, uric acid, Ca, P, serum total cholesterol, high-density lipoprotein cholesterol and triglyceride levels will be measured using standard enzymatic automated methods. Low-density lipoprotein cholesterol will be estimated by the Friedewald equation when the direct parameter is not available. Glycated haemoglobin will be measured with an immune-turbidimetric assay. Cytokines concentrations in plasma will be determined by ELISA using commercial kits and following the manufacturer's recommendations. Oxidative stress will be determined by measuring lipid peroxides and nucleic acid derivatives by ELISA using commercial kits and following the manufacturer's recommendations.
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other:  — No intervention study is an observational study

SUMMARY:
Introduction: The process of population aging that is occurring in developed societies represents a major challenge for the health system. The aim of this study is to analyze factors that have an influence on early vascular aging (EVA), estimated by carotid-femoral pulse wave velocity (cf-PWV) and Cardio Ankle Vascular Index (CAVI), and to determine differences by gender in a Spanish population.

Methods and analysis: An observational, descriptive, cross sectional study.

Study Population: From the population assigned to the participating Health Care centers, a cluster random sampling stratified by age and gender will be performed to obtain 500 participants aged between 35 and 75. Those who meet the inclusion criteria and give written informed consent will be included in the study.

Measurements: Main dependent variables: cf-PWV determined using Sphigmo Cor System and CAVI estimated using VASERA. Secondary dependent variables: telomere length, carotid intima-media thickness, central and peripheral augmentation index, ankle-brachial pulse wave velocity, ankle-brachial index, retinal arteriovenous index, and renal and cardiac organ damage. Independent variables: Lifestyles (physical activity, adherence to mediterranean diet, alcohol and tobacco consumption); psychological factors (depression, anxiety, and chronic stress); inflammatory factors and oxidative stress.

Ethics and dissemination: The study has been approved by the clinical research ethics committee of the healthcare area of Salamanca. All study participants will sign an informed consent to agree to participate in the study in compliance with the Declaration of Helsinki and the WHO standards for observational studies. The results of this study will allow the understanding of the relationship of the different influencing factors and their relative weight in the development of EVA. At least five publications in first-quartile scientific journals are planned.

DETAILED DESCRIPTION:
The general objectives of this study are: To establish reference values for vascular structure and function in the population of Salamanca.

Study design:

A cross-sectional, descriptive observational study. The investigators consider subjects with EVA as those having cf-PWV and/or CAVI values greater than the 75th percentile.

Study setting:

To be implemented in the Research Unit of La Alamedilla Primary Care Center, and on the premises of the Hospital and University of Salamanca of the eight participating groups from the Biomedical Research Institute of Salamanca (IBSAL).

Study population:

It will be the urban population attached to the Health Center of Salamanca. Using a random sampling stratified by age groups (35, 45, 55, 65 and 75 years) and gender, 100 subjects will be selected in each group (50 males and 50 females), aged 35 to 75 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 35 to 75 years who agree to participate in the study and do not meet any of the exclusion criteria.

Exclusion Criteria:

* Subjects who are in terminal condition, who cannot travel to the health centers to undergo the corresponding examinations, and those who do not wish to sign the informed consent.
* Subjects with a history of CVD (ischemic heart disease or stroke, peripheral arterial disease or heart failure), diagnosed renal failure in terminal stages (glomerular filtration rate below 30%), chronic inflammatory disease, or acute inflammatory process in the past three months.
* Patients treated with estrogens, testosterone, or growth hormone.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population It will be the urban population attached to the Health Center of Salamanca. Using a random sampling stratified by age groups (35, 45, 55, 65 and 75 years) and gender, 100 subjects will be selected in each group (50 males and 50 females), aged 35 to 75 years.
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Cardio-ankle vascular index | 2 years
  This parameter will be estimated using Vasera device VS-1500.

SECONDARY OUTCOMES:
Brachial-ankle pulse wave velocity (ba-PWV) | 2 years
  This parameter will be estimated using Vasera device VS-1500.
Ankle-brachial index | 2 years
  This parameter will be estimated using Vasera device VS-1500.
Central augmentation index | 2 years
  This parameter will be estimated using the Sphygmo Cor System.
Carotid Intima Media Thickness | 2 years
  A Sonosite Micromax ultrasound device paired with a 5-10 MHz multifrequency high-resolution linear transducer with Sonocal software.
Evaluation of retinal vessels | 2 years
  Retinography will be performed using a Topcon TRC NW 200 non-mydriatic retinal camera (Topcon Europe B.C., Capelle a/d Ijssel, The Netherlands), obtaining nasal and temporal images centered on the disk.
Adherence to the mediterranean diet | 2 years
  Principal endpoint of alimentation, will be measured using the validated 14-point Mediterranean Diet Adherence Screener.
Objective measure of physical activity | 2 years
  It will be measured using Actigraph GT3X accelerometers.
Self-reported physical activity | 2 years
  It will be measured using the International Physical Activity Questionnaire - Short Form.
Sedentary time | 2 years
  It will be measured using the Questionnaire hours seated (Marshall).
Subjective assessment of physical activity | 2 years
  It will be measured using the Paffenbarger Physical Activity Questionnaire.
Carotid-femoral pulse wave velocity | 2 years
  This parameter will be estimated using the Sphygmo Cor System.

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Primary care Research unit. La Alamedilla health centre, Salamanca
  - Manuel A Gómez Marcos, Salamanca

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Gomez-Marcos MA, Martinez-Salgado C, Gonzalez-Sarmiento R, Hernandez-Rivas JM, Sanchez-Fernandez PL, Recio-Rodriguez JI, Rodriguez-Sanchez E, Garcia-Ortiz L. Association between different risk factors and vascular accelerated ageing (EVA study): study protocol for a cross-sectional, descriptive observational study. BMJ Open. 2016 Jun 7;6(6):e011031. doi: 10.1136/bmjopen-2016-011031. PMID 27267107
- [Derived] Gonzalez Falcon D, Gomez-Sanchez L, Gomez-Sanchez M, Rodriguez-Sanchez E, Tamayo-Morales O, Lugones-Sanchez C, Gonzalez-Sanchez S, Diaz M, Gomez-Marcos MA; en representacion de investigadores del estudio EVA. Evolution of arterial stiffness and association with cardiovascular risk factors in the Spanish population. Follow-up EVA. Med Clin (Barc). 2025 May 9;164(9):461-469. doi: 10.1016/j.medcli.2024.11.008. Epub 2025 Jan 11. English, Spanish. PMID 39800597
- [Derived] Gomez-Sanchez L, Gomez-Sanchez M, Rodriguez-Sanchez E, Lugones-Sanchez C, Tamayo-Morales O, Gonzalez-Sanchez S, de Cabo-Laso A, Garcia-Ortiz L, Gomez-Marcos MA; EVA Investigators. Association of Accelerometer-Measured Sedentary Time and Physical Activity with Arterial Stiffness and Vascular Aging in the General Spanish Population, Analyzed by Sex. Rev Cardiovasc Med. 2023 Nov 17;24(11):318. doi: 10.31083/j.rcm2411318. eCollection 2023 Nov. PMID 39076448
- [Derived] Gomez-Sanchez M, Gomez-Sanchez L, Patino-Alonso C, Recio-Rodriguez JI, Alonso-Dominguez R, Sanchez-Aguadero N, Sanchez CL, Sanchez ER, Garcia-Ortiz L, Gomez-Marcos MA; on behalf EVA investigators. Reference values of central blood pressure and central haemodynamic parameters and their relationship with cardiovascular risk factors in a Spanish population: early vascular ageing study. J Hypertens. 2021 Nov 1;39(11):2147-2156. doi: 10.1097/HJH.0000000000002916. PMID 34343142
- [Derived] Gomez-Sanchez M, Gomez-Sanchez L, Patino-Alonso MC, Alonso-Dominguez R, Sanchez-Aguadero N, Recio-Rodriguez JI, Gonzalez-Sanchez J, Garcia-Ortiz L, Gomez-Marcos MA; EVA group. Relationship of healthy vascular aging with lifestyle and metabolic syndrome in the general Spanish population. The EVA study. Rev Esp Cardiol (Engl Ed). 2021 Oct;74(10):854-861. doi: 10.1016/j.rec.2020.06.040. Epub 2020 Oct 31. English, Spanish. PMID 33132098
- [Derived] Gomez-Sanchez M, Gomez-Sanchez L, Patino-Alonso MC, Cunha PG, Recio-Rodriguez JI, Alonso-Dominguez R, Sanchez-Aguadero N, Rodriguez-Sanchez E, Maderuelo-Fernandez JA, Garcia-Ortiz L, Gomez-Marcos MA; EVA Investigators. Vascular aging and its relationship with lifestyles and other risk factors in the general Spanish population: Early Vascular Ageing Study. J Hypertens. 2020 Jun;38(6):1110-1122. doi: 10.1097/HJH.0000000000002373. PMID 32371801
- [Derived] Gomez-Sanchez M, Patino-Alonso MC, Gomez-Sanchez L, Recio-Rodriguez JI, Rodriguez-Sanchez E, Maderuelo-Fernandez JA, Garcia-Ortiz L, Gomez-Marcos MA; EVA Group. Reference values of arterial stiffness parameters and their association with cardiovascular risk factors in the Spanish population. The EVA Study. Rev Esp Cardiol (Engl Ed). 2020 Jan;73(1):43-52. doi: 10.1016/j.rec.2019.04.016. Epub 2019 Sep 12. English, Spanish. PMID 31521574
- [Derived] Garcia-Ortiz L, Recio-Rodriguez JI, Agudo-Conde C, Maderuelo-Fernandez JA, Patino-Alonso MC, de Cabo-Laso A, Rodriguez-Martin C, Gonzalez-Sanchez J, Rodriguez-Sanchez E, Gomez-Marcos MA; on behalf the EVA Investigators group. Noninvasive validation of central and peripheral augmentation index estimated by a novel wrist-worn tonometer. J Hypertens. 2018 Nov;36(11):2204-2214. doi: 10.1097/HJH.0000000000001806. PMID 29846328